CLINICAL TRIAL: NCT04708353
Title: Effect of Two Different Doses of Oral Pregabalin Premedication for Postoperative Pain Relief After Gynecological Surgeries
Brief Title: Oral Pregabalin Premedication for Postoperative Pain Relief
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Asmaa Mohammed Galal El-Deen, lecturer of anesthesia and surgical intensive care, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 19-11-2020
Record Dates: First submitted 2020-11-23; First posted 2021-01-13 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-09

CONDITIONS: Gynecologic Disease
Keywords: Oral Pregabalin; Postoperative Pain Relief; Gynecological Surgeries
MeSH Terms: conditions — Genital Diseases, Female | interventions — Ascorbic Acid; Focal Adhesion Protein-Tyrosine Kinases; E1A-Associated p300 Protein

STUDY DESIGN:
Intervention Model Description: The patients will be allocated randomly using computer generated randomization table into three equal groups
Who Masked: Participant, Outcomes Assessor
Masking Description: double-blinded ( patient and outcome assessors)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- control group (Placebo Comparator): the patient will receive one placebo capsule (vitamin c) once one hour before the operation.
  Interventions: Drug: placebo capsule (vitamin c)
- Group Pregabalin 150 (Active Comparator): the patient will receive one capsule of pregabalin 150 mg once one hour before the operation
  Interventions: Drug: Group pregabalin 150
- Group Pregabalin 300 (Active Comparator): the patient will receive one capsule of pregabalin 300 mg once one hour before the operation
  Interventions: Drug: Group pregabalin 300

INTERVENTIONS:
Drug: placebo capsule (vitamin c) — the patient will receive one placebo capsule (vitamin c) once one hour before the operation
  Arms: control group
Drug: Group pregabalin 150 — the patient will receive one capsule of pregabalin 150 mg once one hour before the operation
  Other Names: p150
  Arms: Group Pregabalin 150
Drug: Group pregabalin 300 — the patient will receive one capsule of pregabalin 300 mg once one hour before the operation
  Other Names: p300
  Arms: Group Pregabalin 300

SUMMARY:
Pain management after gynecological surgeries is essential for early mobilization of the patient, decrease postoperative complication and hospital stay. The use of opioids is associated with adverse effects such as nausea, vomiting, ileus, pruritus, sedation and respiratory depression.

Previous studies stated that pregabalin has been used to reduce pre-operative anxiety, acute postoperative pain, postoperative opioid requirements, postoperative nausea, vomiting and postoperative delirium. The most effective dose of pregabalin to relief postoperative pain with least side effect is still under trial.

In this study we will compare between two different doses of pregabalin when given as oral premedication in patients undergoing gynecological surgeries under spinal anesthesia regarding postoperative pain in order to reduce opioids consumption and subsequently avoid opioid-related adverse effects.

DETAILED DESCRIPTION:
Postoperative pain, nausea and vomiting continue to be one of the most common and unpleasant complications after surgery. The traditional pain treatment with opioids alone is not adequate any more. To optimize pain treatment and postoperative outcome, new analgesics and new combination of already existing analgesics are searched for.

Pain after gynecological surgery usually severe. Uncontrolled acute post-operative pain is associated with dissatisfaction, post-operative complications and considered as a strong risk factor for development of chronic pain. An enhanced recovery pathway for gynecological surgery must include a strategy to effectively control post-operative pain and allow attainment of other Enhanced Recovery After Surgery (ERAS) targets such as early mobilization and return to oral diet whilst reducing the need for opiates.

Beyond increasing the risk of developing opioid use disorder, perioperative opioid consumption may produce undesirable side effects such as nausea, vomiting, constipation, ileus, pruritus, altered mental status, urinary retention, respiratory complications and increased length of hospital stay. While many of these side effects are frustrating to patient in the immediate postoperative period, the most dangerous effects are those that affect the respiratory system such as opioid-induced respiratory depression (ORD) which consider as a significant cause of brain damage and death in the postoperative period.

Opioid reduction strategies prove useful for decreasing total opioid dose and, in turn, their associated adverse effects. Such strategies may include adjuvant non opioid analgesics such as α-2 agonists, gabapentinoids and N-methyl-D-aspartate receptor agonists as well as local, regional or neuraxial anesthesia and modification of surgical technique where possible for operative patients.

Pregabalin is a new synthetic molecule and a structural derivative of the inhibitory neurotransmitter gamma-amino butyric acid. It is a α2-δ ligand that has analgesic, anticonvulsant, anxiolytic and sleep-modulating activities. Pregabalin binds potently to the α2-δ subunit of calcium channels, resulting in a reduction in the release of several neurotransmitters including glutamate, noradrenaline, serotonin, dopamine and substance P.

Pregabalin could reduce the hyperexcitability of dorsal horn neurons induced by tissue damage; therefore it may be useful in the postsurgical pain prevention.

In 2015, a meta-analysis published in British Medical Journal (BMJ) suggested that pregabalin could improve postoperative analgesia and opioid-related adverse effects namely, vomiting and visual disturbances after surgery. However, the use of the pregabalin for acute postoperative pain is still under trial though widely reported.

ELIGIBILITY:
Inclusion Criteria:

* Physical status: ASA I-II
* BMI ≥ 20kg/m2 & ≤ 35kg/m2,
* Written informed consent from the patient.

Exclusion Criteria:

* Patients with known history of allergy to study drugs,
* Patients on ACE inhibitors, anticonvulsant therapy or any drug interacting with pregabalin,
* Patients on chronic alcohol, opioid, tranquilizer or sedative use,
* Patient with renal impairment or heart failure,
* Pregnant females, Psychological, mental disorders or depression,
* Patients receiving anticoagulants therapy or suspected coagulopathy,
* Patients already on pregbalin or gabapentin therapy.

Ages: 21 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female patients scheduled for benign gynecological surgeries (abdominal hysterectomy, myomectomy, adnexal mass or disturbed ectopic pregnancy) under spinal anesthesia.
Enrollment: 90 (Estimated)
Dates: Start 2020-08-20 (Actual); Primary Completion 2021-10 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
changes in Postoperative pain | at 2, 4, 6, 8, 10, 12, 16, 20 and 24 hours postoperatively
  will be assessed by visual analogue scale (VAS), On a scale of 0-10, the patient will learn to quantify postoperative pain where 0= No pain and 10= Maximum worst pain.

SECONDARY OUTCOMES:
The level of sedation | at 2, 4, 6, 8, 10, 12, 16, 20 and 24 hours postoperatively
  using the modified Ramsay Sedation Score:
  1. Patient is anxious and agitated or restless, or both.
  2. Patient is cooperative, oriented and tranquil.
  3. Patient responds to commands only.
  4. Patient exhibits brisk response to light glabellar tap or loud auditory stimulus.
  5. Patient exhibits sluggish response to light glabellar tap or loud auditory stimulus.
  6. Patient exhibits no response.
Total amount of rescue analgesic | in the first 24 hours
  Total amount of rescue analgesic requirement by the patient

CONTACTS AND LOCATIONS:
Locations (1):
- faculty of medicine, Zagazig university, Zagazig, Elsharqya, Egypt

IPD SHARING:
Plan to Share IPD: Yes
planned after the completion of the study and publication
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: planned after the completion of the study and publication
Access Criteria: principal investigator

REFERENCES:
- [Background] Guay DR. Pregabalin in neuropathic pain: a more "pharmaceutically elegant" gabapentin? Am J Geriatr Pharmacother. 2005 Dec;3(4):274-87. PMID 16503325
- [Background] Dahl JB, Mathiesen O, Moiniche S. 'Protective premedication': an option with gabapentin and related drugs? A review of gabapentin and pregabalin in in the treatment of post-operative pain. Acta Anaesthesiol Scand. 2004 Oct;48(9):1130-6. doi: 10.1111/j.1399-6576.2004.00484.x. PMID 15352959
- [Background] Mishriky BM, Waldron NH, Habib AS. Impact of pregabalin on acute and persistent postoperative pain: a systematic review and meta-analysis. Br J Anaesth. 2015 Jan;114(1):10-31. doi: 10.1093/bja/aeu293. Epub 2014 Sep 10. PMID 25209095
- [Background] Balaban F, Yagar S, Ozgok A, Koc M, Gullapoglu H. A randomized, placebo-controlled study of pregabalin for postoperative pain intensity after laparoscopic cholecystectomy. J Clin Anesth. 2012 May;24(3):175-8. doi: 10.1016/j.jclinane.2011.06.027. Epub 2012 Mar 28. PMID 22459341